CLINICAL TRIAL: NCT04893330
Title: Interest of Peticate Syneo Infant Formula in Children Allergic to Cow's Milk Protein: Real Life Study
Acronym: PEPSY
Status: Completed | Type: Observational
Sponsor: Nutricia Nutrition Clinique (Industry)
Responsible Party: Sponsor
Other Study IDs: 2021- A00703-38
Record Dates: First submitted 2021-05-07; First posted 2021-05-19 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2022-04

CONDITIONS: Milk Hypersensitivity
MeSH Terms: conditions — Milk Hypersensitivity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients: children under 8 months of age at inclusion, with a diagnosis or strong suspicion of APLV
  Interventions: Dietary Supplement: pepticate syneo

INTERVENTIONS:
Dietary Supplement: pepticate syneo — follow up of pepticate syneo for one month

SUMMARY:
Nutricia wants to launch a real-life study, to see how the presence of prebiotics and probiotics in the boosted protein hydrolyzate can improve symptoms in the first weeks of use, and supplement the efficacy and safety data of the drug. formula, collected during clinical trials, with real life use. The target population will be children with a definite or suspected diagnosis of APLV, who have never taken a hypoallergenic formula, for whom the doctor decides to prescribe the Pepsicate Syneo formula, regardless of the clinical manifestation of the allergy. These children will be included before the age of 8 months and will be seen again 4 weeks after the prescription. The data from this real-life study will also better characterize the profile of infants taking Pepsicate Syneo. Finally, the perception of the formula by the parents will be collected.

DETAILED DESCRIPTION:
Nutricia has developed an infant formula intended for children, APLV, from the class of foodstuffs intended for special medical purposes (DADFMS), called Pepticate Syneo. This hypoallergenic formula is based on high hydrolyzate of whey protein. It also contains:

* IcFOS and scGOS prebiotic fibers. These oligosaccharides are well tolerated and promote the induction of a favorable gut microbiota and an improvement in faecal characteristics [Arslanoglu 2008, Moro 2006].
* The probiotic strain Bifidobaterium Breve M-16V. B. breve is the most common species of bifidobacteria in human milk [Martin 2009]. The B. breve M16-V strain, isolated from the stool of a healthy infant, is approved in food by health authorities and conforms to the recommendations of the American Academy of Pediatrics [2000]. It helps promote the implantation of beneficial bacteria in the intestinal microbiota of young children [Akiyama 1994, Taniuchi 2005, van der Aa 2010]. Preclinical data suggest that it reduces the allergic immune response [Hougee 2010, Inoue 2009]. In clinical studies, it helps reduce atopic dermatitis in children with APLV [Hattori 2003, Taniuchi 2005]. In addition, the prebiotic / probiotic combination (also called symbiotic) shows a synergistic effect in mice in reducing allergic manifestations [Schouten 2009]. Used in children born by cesarean section, it helps restore intestinal colonization by bifidobacteria, to a level similar to that of infants born vaginally and breastfed [Chua 2017].

In babies with a suspicion of non-IgE-mediated APLV, this symbiotic mixture (IcFOS, scGOS and B. Breve) allowed a modification of the fecal microbiota in 8 weeks, thus approaching the microbiota of breastfed infants of the same age, with an increase in Bifidobacteria and a decrease in Eubacterium rectale / Clostridium coccoides [Fox 2019].

All the available scientific data suggest an excellent tolerance of the Pepticate Syneo formula, and therapeutic efficacy on the manifestations of APLV, whether or not it is mediated by IgE, while ensuring the nutritional needs of children's growth. [Abrahamse-Berkeveld 2016, Giampietro 2001, Vandenplas 1993, Verwimp 1995].

ELIGIBILITY:
Inclusion Criteria:

* Child aged ≤ 8 months;
* Child newly diagnosed with an allergy to cow's milk proteins (APLV), or with a strong suspicion of APLV (mediated by IgE or not), justifying (according to the doctor) the prescription of Pepticate® Syneo® (extensive hydrolyzate cow's milk protein)
* Child already fed with an infant formula (partially or totally), or whose parents have already made the decision to initiate an infant formula, in addition to or as a follow-up to breastfeeding.
* Authorization of one or more parents or the child's legal representative to collect personal information about the child and the family.

Exclusion Criteria:

* Child who has already taken an infant formula such as "high protein hydrolyzate" or "amino acid formula";
* Child with a contraindication to taking symbiotics (eg: short bowel syndrome, parenteral nutrition, post-pyloric nutrition, central venous catheter, etc.)
* Child with severe APLV requiring the prescription of an amino acid formula;
* Legal guardian of the protected child (under legal protection, or deprived of liberty by judicial or administrative decision);
* Legal guardian of the child who is not a beneficiary of a social security scheme.
* Inability of the legal representative to understand the study protocol, or doctor's doubts about the ability of the will to comply with the protocol.

Min Age: 8 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The target population is made up of children under 8 months of age at inclusion, with a diagnosis or strong suspicion of APLV.
  The study plans to include 78 patients.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2021-06-23 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
effect on general condition | Day 28
  Assessment of the effect of the PEPTICATE SYNEO formula on the evolution of the general condition of a child with a PPLA using a 4-level Likert scale (worse / identical / improved / resolved)

SECONDARY OUTCOMES:
Effect on evolution of allergic symptoms | Day 28
  Evaluation of the effect of the PEPTICATE SYNEO formula on the evolution of allergy symptoms using a 4-level Likert scale (worse / identical / improved / resolved)
effect on evolution of allergic symptoms according to Parents | during one month
  Assessment of the effect of the PEPTICATE SYNEO formula on the evolution of allergy symptoms according to the parents using a 4-level Likert scale (worse / identical / improved / resolved)
acceptability | Day 28
  Descriptive analysis of the acceptability of PEPTICATE SYNEO by parents using a questionnaire
Parent's quality of life | Day 28
  The quality of life of the parents (FAQL-PB score) will be measured by a Student test on paired samples.
CLINICAL PROFILE OF CHILDREN | Day 0
  Description of the clinical profile of the children at inclusion (Age, anthropometric data; growth; Food history, Risk factors for atopy..).
Consumption of the formula | during one month
  Evaluation of the infant formula consumption of children before inclusion and during follow-up (lasting 28 days).

CONTACTS AND LOCATIONS:
Locations (1):
- Cabinet Médical, Charly, France

IPD SHARING:
Plan to Share IPD: No